CLINICAL TRIAL: NCT06154707
Title: Clinical Controlled Study on the Efficacy of Denosumab in Treating Osteoporosis in the Domestic Population and Its Impact on Sarcopenia-related Outcomes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHCT230847
Record Dates: First submitted 2023-11-10; First posted 2023-12-04 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia; Osteoporosis; Denosumab
MeSH Terms: conditions — Sarcopenia; Osteoporosis | interventions — Denosumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab Group (Experimental): Denosumab injection 60mg (1.0ml/ branch, Jiangsu Taikang Biological Medicine Co., LTD., s20233111), once every 6 months, 60mg, subcutaneous injection, at the same time to supplement calcium and vitamin D.
  Interventions: Drug: Denosumab Injection
- Placebo Group (Placebo Comparator): Placebo drug, the main component of normal saline injection (1.0ml/ dose). In addition to the different production batch number, its appearance, character, specification, administration mode and frequency are exactly the same as the experimental group of drugs (different production batch number is convenient for later unblinding reference). Take calcium and vitamin D supplements. The study lasted for 12 months.
  Interventions: Other: Normal saline injection (1.0ml/ branch)

INTERVENTIONS:
Drug: Denosumab Injection — Denosumab injection 60mg (1.0ml/ branch, Jiangsu Taikang Biological Medicine Co., LTD., s20233111), once every 6 months, 60mg, subcutaneous injection, at the same time to supplement calcium and vitamin D.
  Arms: Denosumab Group
Other: Normal saline injection (1.0ml/ branch) — Placebo drug, the main component of normal saline injection (1.0ml/ dose). In addition to the different production batch number, its appearance, character, specification, administration mode and frequency are exactly the same as the experimental group of drugs (different production batch number is convenient for later unblinding reference). Take calcium and vitamin D supplements.
  Arms: Placebo Group

SUMMARY:
Through the method of a clinical randomized controlled trial, patients meeting the study criteria are randomly assigned to either the Denosumab treatment group or a placebo group. After a treatment period of 12 months, the differences in osteoporosis and sarcopenia-related baseline assessment changes between the two groups are compared. This is to explore the effect of Denosumab in treating osteoporosis and its impact on sarcopenia. The goal is to evaluate the efficacy of Denosumab in treating osteoporosis in the domestic population and its related impact on sarcopenia, with the aim of providing an effective treatment option for the domestic population suffering from 'osteoporosis-sarcopenia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of postmenopausal/senile osteoporosis after examination and assessment.
* Clinical diagnosis of postmenopausal/senile osteoporosis combined with sarcopenia after examination and assessment.
* Have not previously taken any other anti-osteoporosis drugs.

Exclusion Criteria:

* Clinical diagnosis of pathological fractures.
* Have participated in another clinical trial within the past 3 months or have taken other anti-osteoporosis drugs within the past 6 months.
* Severe chronic metabolic diseases or serious organ failure.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis-related Primary Outcome | 1 year
  Bone mineral density (BMD) changed from baseline after 6 and 12 months of treatment in both groups. (DXA method, T value has no specific unit of measure)
  Bone transformation markers (BTM) changed from baseline after 6 and 12 months of treatment in both groups. (Total P1NP（ng/ml）, total 25 hydroxyvitamin D（nmol/L）, osteocalcin N-terminal fragment（ng/ml）, βCrossLap（pg/ml）)
  After 6 and 12 months of treatment, osteoporosis related blood biochemistry(TBIL, DBIL, Cr, UA, HCY in umol/L, BUN, TC, TG, HDL, LDL, Ca, IP in mmol/L, ALB, PAB in g/L, CK, ALT, AST, GGT in U/L), blood routine(WBC, PLT, NEU, LYMPH, MONO, EOS in G/L, RBC in T/L, HGB in g/L), inflammatory indicators(IL-1β, TNF-α, IL-6 in pg/mL), and related hormones(PTH, CT in ng/L) changed from baseline.
  Changes in the above indicators from the baseline are possible or hypothetical, and all are subject to experimental results.
Sarcopenia-related Primary Outcome | 1 year
  After 6 and 12 months of treatment, the SARC-F scale was evaluated compared with baseline.(No unit of measure)
  After 6 and 12 months of treatment, muscle strength (dominant hand grip strength, Kg) changed from baseline in both groups.
  After 6 and 12 months of treatment, skeletal muscle mass (ASM in Kg), skeletal muscle mass index (ASM and height will be combined to report ASMI in Kg/m²), body fat percentage（%） and limb fat percentage（%）in both groups were changed from baseline. (BIA method)
  After 6 and 12 months of treatment, the walking speed of 6 M（m/s） and the sitting time of 5 times(s) were changed from baseline.
  Changes in the above indicators from the baseline are possible or hypothetical, and all are subject to experimental results.

SECONDARY OUTCOMES:
Quality of life and fall risk | 1 year
  Changes in quality of life and fall risk from baseline were assessed using the abbreviated Health Survey Form (SF-36) and the Morse Fall Risk Assessment Scale at the end of 12 months of treatment in both groups.(The score has no specific unit of measure)
  Changes in the above scale from the baseline are possible or hypothetical, and all are subject to experimental results.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China